CLINICAL TRIAL: NCT00453583
Title: Evaluation of the Treatment Satisfaction in Children Suffering From an Allergy and Who Received an Antihistamine Treatment
Brief Title: Evaluation of Treatment Satisfaction in Children With an Allergy and Who Received an Antihistamine
Status: Completed | Type: Observational
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: A00420
Record Dates: First submitted 2007-03-28; First posted 2007-03-29 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2012-05

CONDITIONS: Allergies
Keywords: Pediatric; Allergies; Antihistamines; Non-interventional
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
This is a non-interventional retrospective data collection study from children aged from 2 to 12 years old diagnosed with an allergy and who received a treatment consisting of an H1-antihistamine. The period of last taken medication will be observed to evaluate the global satisfaction of the parents and physician for this last treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children from 2-12 included
* History of allergy
* Used an Antihistamine within market authorization

Exclusion Criteria:

* Child not yet treated for the presented allergy

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Primary Care
Sampling Method: Non-Probability Sample
Enrollment: 4581 (Actual)
Dates: Start 2007-03; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Parent satisfaction on a 11-point scale | duration of the study

SECONDARY OUTCOMES:
Physician satisfaction on an 11-point scale | duration of the study
Efficacy, tolerability and global satisfaction | duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- UCB Pharma, Smyrna, Georgia, United States